CLINICAL TRIAL: NCT04887012
Title: Clinical Study of HLA Haploidentical CAR-NK Cells Targeting CD19 in the Treatment of Refractory/Relapsed B-cell NHL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2021002168
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK019 (Experimental): All subjects were intravenously administrated with CAR-NK019
  Interventions: Biological: anti-CD19 CAR-NK

INTERVENTIONS:
Biological: anti-CD19 CAR-NK — lentiviral vector-transducted HLA haploidentical NK cells to express anti-CD19 CAR
  Other Names: CAR-NK019

SUMMARY:
To study the safety and effectiveness of HLA haploidentical CAR-NK cells targeting CD19 in patients with B-cell non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study and sign an informed consent form;
2. Age 18-75 years old, no gender limit;
3. Histologically diagnosed as diffuse large B-cell lymphoma (DLBCL), transforming follicular lymphoma (TFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL) and other inert B-cells NHL conversion type:

   * Refractory or relapsed DLBCL refers to the failure to achieve complete remission after 2-line treatment; disease progression during any treatment, or disease stable time equal to or less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation ；
   * Refractory or relapsed MCL must be resistant to or intolerable to BTK inhibitors;
   * Refractory or relapsed indolent B-cell NHL is the failure or recurrence of third-line treatment;
   * Previous treatment must include CD20 monoclonal antibody treatment (unless the subject is CD20 negative) and anthracyclines;
4. At least one measurable lesion with the longest diameter ≥ 1.5 cm exists;
5. The expected survival period is ≥12 weeks;
6. The puncture section of the tumor tissue was positive for CD19 expression;
7. ECOG score 0-2 points;
8. Sufficient organ function reserve:

   * Alanine aminotransferase, aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value);
   * Creatinine clearance rate (Cockcroft-Gault method) ≥60 mL/min;
   * Serum total bilirubin and alkaline phosphatase ≤1.5× UNL;
   * Glomerular filtration rate>50Ml/min
   * Cardiac ejection fraction (EF) ≥50%;
   * Under natural indoor air environment, basic oxygen saturation>92%
9. Allow a previous stem cell transplantation
10. The approved anti-B-cell lymphoma treatments, such as systemic chemotherapy, systemic radiotherapy, and immunotherapy, have been completed for at least 3 weeks before the study medication;
11. Allow patients who have previously received CAR-T cell therapy and have failed or relapsed after 3 months of evaluation;
12. Female subjects of childbearing age must have a negative pregnancy test and agree to take effective contraceptive measures during the trial
13. Two tests for the new coronavirus were negative.

Exclusion Criteria:

1. Those who have a history of allergies to any of the ingredients in cell products;
2. History of other tumors
3. Previously presented with II-IV degree (Glucksberg criteria) acute GvHD or extensive chronic GvHD; or are receiving anti-GvHD treatment;
4. Have received gene therapy in the past 3 months;
5. Active infections that require treatment (except for simple urinary tract infections and bacterial pharyngitis), but preventive antibiotics, antiviral and antifungal infection treatments are allowed;
6. Hepatitis B (HBsAg positive, but HBV-DNA <103 is not an exclusion criterion) or hepatitis C virus infection (including virus carriers), syphilis and other subjects with acquired and congenital immunodeficiency diseases, including But not limited to people living with HIV;
7. According to the New York Heart Association's Heart Function Classification Standard, it is classified as Grade III or Grade IV.

   Impaired subjects;
8. Those who have received anti-tumor therapy in the early stage but the toxic reaction has not recovered (the CTCAE 5.0 toxic reaction has not recovered to ≤1, except for fatigue, anorexia, and hair loss);
9. Subjects with a history of epilepsy or other central nervous system diseases;
10. Enhanced CT or MRI of the head showed evidence of central nervous system lymphoma;
11. Have received any other drugs that target CD19;
12. Women who are breastfeeding and unwilling to stop breastfeeding;
13. Any other situation that the investigator believes may increase the risk of the subject or interfere with the results of the test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of Anti-CD19 CAR-NK Cell Therapy for B-cell Non-Hodgkin Lymphoma
The overall response rate(ORR) | Up to 2 years
  To determine the anti-tumor effectivity of CAR-NK019

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of CAR-NK019
progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of CAR-NK019
Pharmacokinetics of CAR positive cells | Up to 2 years
  The copy number of CAR DNA was measured at the preset follow-up time point.
Pharmacokinetics of CAR-NK cells | Up to 2 years
  The duration of CAR-positive NK cells in circulation was measured by FACs

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No